CLINICAL TRIAL: NCT03125148
Title: Comparison of Duodenal Stenting vs Transpyloric and Duodenal Stenting for Malignant Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Kulwinder Dua, MD, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00028657
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Duodenal Obstruction
MeSH Terms: conditions — Duodenal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Enteral stenting intraduodenal (Active Comparator): Enteral stent (Wallflex enteral stent) will be placed in the duodenum with the entire stent lying within the duodenum bridging the obstruction.
  Interventions: Device: Enteral stenting
- Enteral stenting transpyloric (Experimental): Enteral stent (Wallflex enteral stent) will be placed in the duodenum with the stent bridging the obstruction and the pyloric opening with proximal end of the stent lying within the stomach
  Interventions: Device: Enteral stenting

INTERVENTIONS:
Device: Enteral stenting — Enteral stent for malignant duodenal obstruction

SUMMARY:
Malignant duodenal obstruction in patients not fit for surgery is treated by placing enteral stents during endoscopy. These patients may also have poor gastric motility. Hence bridging the pyloric opening with the stent along with the duodenal obstruction may deliver better symptomatic improvement. Both approaches are commonly clinically practiced but no formal comparative studies have been done to compare which one is better.

DETAILED DESCRIPTION:
Enteral self-expanding metal stents are routinely used to palliate malignant gastric outlet obstruction (pancreas cancer, duodenal cancer, gastric cancer and metastasis) in patients not fit for surgical bypass. The technical success in placing these stents approaches ~100% and many of these procedures can be performed in an outpatient setting. However the functional success (patient's ability to eat) is much lower than the technical success. One of the major reasons for this discrepancy is these patients are on narcotics, which are known to be associated with poor gastric motility. At the discretion of the gastroenterologist, FDA approved enteral stents are placed either completely within the duodenum bridging the obstruction or placed across the pyloric opening besides bridging the duodenal obstruction. The significance of this study is to determine if trans-pyloric extension of an intra-duodenal stent facilitates better gastric emptying compared to an intra-duodenal stent without trans-pyloric extension.

ELIGIBILITY:
Inclusion Criteria:

1 - Confirmed diagnosis of cancer

2. Evidence of a single small bowel obstruction

3. Considered palliative (can be on narcotics, chemotherapy, and/or radiation therapy)

4. Not a surgical candidate

5. >18 years of age

6. Able to give consent

7. Eligible for endoscopy (medically fit)

8. Able to traverse past obstruction with a guidewire

Exclusion Criteria:

1 - <18 years of age

2. Unable to give consent

3. Pregnant

4. Have evidence of multiple sites of obstruction in the small bowel

5. Have evidence of duodenal obstruction secondary to gastric cancer

6. Ineligible for endoscopy (due to comorbidities or acuity of illness)

7. Unable to traverse past obstruction with a guidewire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rusch, PhD, Study Chair — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enteral Stenting Intraduodenal: GROUP A: Enteral stent (Wallflex enteral stent) will be placed in the duodenum with the entire stent lying within the duodenum bridging the obstruction.
  Enteral stenting: Enteral stent for malignant duodenal obstruction
- Enteral Stenting Transpyloric: GROUP B: Enteral stent (Wallflex enteral stent) will be placed in the duodenum with the stent bridging the obstruction and the pyloric opening with proximal end of the stent lying within the stomach
  Enteral stenting: Enteral stent for malignant duodenal obstruction
Period: Overall Study
Arm/Group | Enteral Stenting Intraduodenal | Enteral Stenting Transpyloric
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteral Stenting Intraduodenal | Enteral Stenting Transpyloric | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Change (2 Point Increase or Decrease) in Symptoms From Baseline
Description: Symptoms of nausea, regurgitation, bloating, fullness, belching, pain, and vomiting were recorded at baseline and then on follow-up after stent placement on a visual analog scale with 0 being no symptoms and 10 being severe symptoms. The visual analog scale used was: 0 No symptom to 10 Severe symptom: Drop by 2 points or more from baseline score after intervention was recorded as "Better" and increase in over 2 points from baseline after intervention was recorded as symptom getting "Worse". A -1 to +1 shift from baseline was considered as "Unchanged".
  Gastric emptying was objectively assessed at 48 hours after stent placement with no baseline testing.
  Over all quality of life change after stent placement over baseline was a subjective response from the patient as being "Satisfied", "Neutral", "Dissatisfied." Re-interventions and adverse events if any were recorded.
Time Frame: Baseline (before stent) and follow-up (after stent) at 48 hrs (including gastric emptying study) and then symptom follow up at each clinic/telephone visit up to 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Stenting Intraduodenal | Enteral Stenting Transpyloric
Number analyzed (Participants) | 9 | 8
Participants | 7 | 6

2. Secondary Outcome: Technical Success: Stent Placed in the Desired Position as Per Randomization
Description: Successful placement of the stent across the duodenal obstruction with or without trans-pyloric extension as per randomization will determined immediately during endoscopic procedure by endoscopic visualization.
Time Frame: Day of stent deployment
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Stenting Intraduodenal | Enteral Stenting Transpyloric
Number analyzed (Participants) | 9 | 8
Participants | 9 | 8

3. Secondary Outcome: Complications
Description: Stent related complications
Time Frame: Up to 6 months after stent deployment
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Stenting Intraduodenal | Enteral Stenting Transpyloric
Number analyzed (Participants) | 9 | 8
Participants | 0 | 0

4. Secondary Outcome: Gastric Emptying
Description: Gastric emptying study test
Time Frame: 48 hours after stent placement
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral Stenting Intraduodenal | Enteral Stenting Transpyloric
Number analyzed (Participants) | 9 | 8
Participants | 5 | 2

ADVERSE EVENTS:
Time Frame: Median 29 days Range 7-462 days
Arm/Group | Enteral Stenting Intraduodenal | Enteral Stenting Transpyloric
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT03125148/Prot_SAP_001.pdf